CLINICAL TRIAL: NCT04329455
Title: Evaluation of Endoscopic Thyroidectomy Via Axillo-breast Approach in Thyroid Nodules
Acronym: Thyroidectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Hemdan, MD, Assiut University
Other Study IDs: Ahmed1989
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Safety and Cosmetic Issues in Endoscopic Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention group
  Interventions: Procedure: Endoscopic thyroidectomy

INTERVENTIONS:
Procedure: Endoscopic thyroidectomy — Endoscopic thyroidectomy in Thyroid Nodules

SUMMARY:
Evaluation of Endoscopic Thyroidectomy via Axillo-breast Approach in Thyroid Nodules regarding safety and cosmetic outcomes

ELIGIBILITY:
Inclusion Criteria:

* benign thyroid nodules unilateral or bilateral Normal thyroid function

Exclusion Criteria:

* malignant Thyroid Nodules Recurrent goitre Toxic goitre

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 patients age group 18_55 years with unilateral or bilateral thyroid nodules benign according to preoperative FNAC and normal thyroid function
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Endoscopic Thyroidectomy | 2020_2023

SECONDARY OUTCOMES:
Cosmetic outcome of Endoscopic Thyroidectomy | 2020_2023

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Gamal, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No